CLINICAL TRIAL: NCT03551340
Title: Impact of the Introduction of a Gastro-intestinal Panel by PCR on the Treatment of Patients With Gastroenteritis
Brief Title: Impact of the Introduction of a Gastro-intestinal Panel by Polymerase Chain Reaction (PCR).
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Serge de Valliere, PD & MER, University of Lausanne Hospitals
Other Study IDs: 2017-02042
Record Dates: First submitted 2018-05-28; First posted 2018-06-11 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Gastroenteritis
Keywords: Gastroenteritis, panel by PCR, antibiotic use
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Traditional methods: Patients, who consulted for gastro-intestinal symptoms between July 2016 and May 2017, and were investigated by traditional methods (stool microscopy and/or culture).
- Gastro-intestinal panel by PCR: Patients, who consulted for gastro-intestinal symptoms between July 2017 and May 2018,and were investigated by a gastro-intestinal panel by PCR
  Interventions: Diagnostic Test: Gastro-intestinal panel by PCR

INTERVENTIONS:
Diagnostic Test: Gastro-intestinal panel by PCR — The study will evaluate the change in medical management with the replacement of traditional stool investigations (microscopy and culture) by the new gastrointestinal multiplex PCR panels
  Groups: Gastro-intestinal panel by PCR

SUMMARY:
Evaluation of the impact of the introduction of multiplex PCR panels on the clinical management of patients with gastroenteritis at the University Hospital of Lausanne, Switzerland.

DETAILED DESCRIPTION:
Gastrointestinal multiplex PCR panels have been introduced in clinical practice several years ago, but the impact on the management of patients is yet unknown. The investigators are interested to evaluate if the multiplex PCR panels introduced at the University Hospital of Lausanne in July 2017 modified the usual medical care and in particular the prescription of anti-infectious treatments. The high sensitivity of the multiplex PCR panels should allow a more precise diagnosis of the etiology of the gastrointestinal symptoms of the patients than the traditional methods of stool culture and microscopy. The investigators expect therefore to observe a modification of the proportion of patients receiving anti-infectious treatment, but it is uncertain if it will lead to an increase or a decrease in the use of antibiotics. On one hand antibiotics could be prescribed more often due to a greater and faster detection of enteropathogens. On the other hand antibiotics could be prescribed less often due to more precise diagnosis, showing that viruses and certain bacteria do not require antibiotic treatment.

ELIGIBILITY:
Inclusion criteria:

Ambulatory patients who consulted the University Hospital of Lausanne between July 2016 and May 2017, and were investigated by traditional methods (stool microscopy and culture).

Ambulatory patients who consulted the University Hospital of Lausanne between July 2017 and May 2018 and had stool investigations by a gastro-intestinal panel.

Exclusion criteria:

Patients for whom there ia record in the file that they do not accept that their data are used for research purposes.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulting the emergency department of the University Hospital of Lausanne for gastro-intestinal symptoms suggestive of an infectious origin
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Prescription of antibiotics | Within 1 week of availability of stool result
  Number of patients receiving a prescription of antibiotics depending on the type of investigation

SECONDARY OUTCOMES:
Pathogens identified | 1 day
  Number and types of pathogens identified depending on the type of investigation
Number of PCR tests requested. | 1 month
  Number of patients for whom one, two or more PCR tests were requested.
Additional investigations | 1 week
  Number of patients who underwent additional investigations within 1 week after reception of the results of the initial investigations

CONTACTS AND LOCATIONS:
Overall Officials: Serge de Valliere, MD,MSc, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Department of Outpatient Care and Community Medicine, University Hospital of Lausanne, Lausanne, Switzerland